CLINICAL TRIAL: NCT07390318
Title: Comparing Antegrade Versus Retrograde Enemas To Improve Bowel Continence Across the Lifespan in People With Spina Bifida
Brief Title: Bowel Continence Across the Lifespan in People With Spina Bifida
Acronym: BCALS
Status: Not yet recruiting | Type: Observational
Sponsor: David Chu (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor-Investigator, David Chu, Principal Investigator; Attending Physician, Urology; Associate Professor of Urology at Northwestern University Feinberg School of Medicine, Ann & Robert H Lurie Children's Hospital of Chicago
Organization: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Other Study IDs: STUDY00000320
Record Dates: First submitted 2026-01-28; First posted 2026-02-05 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Spina Bifida; Neurogenic Bowel; Bowel Incontinence
Keywords: retrograde enema; antegrade enema; bowel management program; bowel continence program; self-management; quality of life
MeSH Terms: conditions — Spinal Dysraphism; Neurogenic Bowel; Fecal Incontinence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Retrograde Enema: Participants starting a retrograde enema program, as part of standard care prescribed by their local clinical team.
  Interventions: Procedure: Retrograde Enema
- Antegrade Enema: Participants starting an antegrade enema program, as part of standard care prescribed by their local clinical team.
  Interventions: Procedure: Antegrade Enema

INTERVENTIONS:
Procedure: Retrograde Enema — A retrograde enema is a bowel management technique in which the enema is given through the rectum (end of the colon). This includes cone enemas, foley balloon enemas, and Transanal irrigation (e.g. Peristeen, Navina).
  Groups: Retrograde Enema
Procedure: Antegrade Enema — An antegrade enema is a bowel management technique in which an enema is given through a surgically-created tube that enters at the start of the colon. This includes MACES, cecostomy buttons, and Chait tubes.
  Groups: Antegrade Enema

SUMMARY:
The goal of this observational study is to learn how different enema programs affect bowel control in children and adults with spina bifida. An enema program involves putting liquid into the large intestine (colon) to help someone poop. The main questions it aims to answer are:

1. How well do different enema programs prevent bowel accidents?
2. How do these enema programs affect independence, bowel symptoms, and quality of life?

Researchers will compare two types of enema programs to see which works better and is easier for participants to manage.

Participants starting a new enema program will answer online survey questions at 3 different timepoints over the course of 1 year.

DETAILED DESCRIPTION:
Spina bifida is a rare disease affecting an estimated 166,000 people in the United States. Because of the birth defect in the spinal cord, many organ systems do not work properly. Included among these affected organ systems are the bowels or intestines, which can lead to bowel incontinence or bowel accidents. Bowel incontinence is very disruptive to the lives of people with spina bifida by affecting their ability to have romantic relationships, find jobs, and overall enjoy their lives. The spina bifida community has recognized bowel incontinence as a top priority for research.

Typically, reducing bowel incontinence and improving bowel continence occurs in a stepwise fashion. After medications by mouth such as laxatives or stool softeners, 2nd line treatments include enema programs. Two types of enema programs currently exist, those given in either a backward direction (given through the anus or end of the large intestine or colon) or in a forward direction (given through a tube that enters the start of the large intestine or colon). These two types of enema programs have different positives and negatives which have not been compared nor studied well. The lack of evidence on which is the better enema program presents a key decisional dilemma for many people with spina bifida who want to improve their bowel continence.

In the current study, the study team will compare the two types of enema programs in 943 children and adults ages 5 years old and up with spina bifida at 24 centers across the United States. The enema programs will be assigned to and started by the participants as part of usual clinical care from their local clinical team. At 6 months and 12 months over a 1-year study period, the study team will look at how the two types of enema programs compare in bowel continence (how well they work to prevent bowel accidents), quality of life (how much people enjoy their lives), bowel symptoms (how well they work to reduce bowel-related symptoms), self-management and independence (how well people can do these enema programs themselves without help), and healthcare utilization (how often these enema programs cause problems needing medical help). The study team will also ask 20 children with spina bifida, 20 adults with spina bifida, and 20 caregivers of children and adults with spina bifida more detailed interview questions about their lived experiences with managing bowel incontinence and their thoughts on how best to start and maintain a successful enema program. The expected study results will help people with spina bifida not only improve their bowel continence, but also their quality of life.

The study team is working with patient and family partners within the spina bifida community, healthcare providers across numerous disciplines, national advocacy organizations (the Spina Bifida Association), and industry partners who make enema devices to design and conduct this study.

ELIGIBILITY:
Inclusion Criteria:

* Minimum age 5 years old
* Myelomeningocele diagnosis
* Starting a retrograde or antegrade enema program (or switching from one enema program to the other)
* English or Spanish speaking/literate

Exclusion Criteria:

- Other types of spinal dysraphism (e.g., lipomyelomeningocele, fatty filum)

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Children, adolescents, and adults age 5 years and older with spina bifida starting a new enema program at one of 24 participating clinical centers in the United States.
Sampling Method: Non-Probability Sample
Enrollment: 943 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2030-05-01 (Estimated); Study Completion 2030-05-01 (Estimated)

PRIMARY OUTCOMES:
Bowel continence | Before starting enema program, 6 months after starting enema program, 1 year after starting enema program
  Measured with a single question on bowel incontinence frequency in the past month, with "continence" strictly defined as answering "never": (Daily, Weekly, Monthly, Never)

SECONDARY OUTCOMES:
Bowel symptoms and satisfaction | Before starting enema program, 6 months after starting enema program, 1 year after starting enema program
  Measured using the Neurogenic Bowel Dysfunction (NBD) score. Scores range from 0-47, higher scores mean greater severity of bowel dysfunction.
Disease-specific quality of life | Before starting enema program, 6 months after starting enema program, 1 year after starting enema program
  Measured using the Quality of Life Assessment in Spina Bifida (QUALAS) Child, Teenager, and Adult questionnaires. Scores range from 0-100, higher scores mean better quality of life.
Overall quality of life | Before starting enema program, 6 months after starting enema program, 1 year after starting enema program.
  Measured using the Patient-Reported Outcomes Measurement Information System (PROMIS) Global Health and Pediatric Global Health 7 questionnaires. Raw scores are converted into T-scores, which range from 16.2-67.7 for PROMIS Global Health and 16-67.5 for PROMIS Pediatric Global Health 7. Higher scores mean better quality of life.
Self-management and independence | Before starting enema program, 6 months after starting enema program, 1 year after starting enema program
  Measured using the Adolescent/Young Adult Self-Management and Independence Scale (AMIS) II. Scores range from 36-252, higher scores mean higher level of self-management and independence.
Rate of unplanned healthcare utilization related to bowel issues | For 1 year after starting enema program
  Number of emergency room visits, urgent care or immediate care visits, and urgent outpatient ambulatory visits related to bowel issues.

CONTACTS AND LOCATIONS:
Locations (24):
- United States (24):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Children's of Alabama, Birmingham, Alabama
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Children's Hospital of Los Angeles, Los Angeles, California
  - University of California San Francisco, San Francisco, California
  - Children's Hospital of Colorado, Denver, Colorado
  - Children's National Hospital, Washington D.C., District of Columbia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Northwestern University, Chicago, Illinois
  - Riley Children's Hospital, Indianapolis, Indiana
  - Boston Children's Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Duke University Medical Center, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Monroe Carell Jr. Children's Hospital at Vanderbilt, Nashville, Tennessee
  - Scottish Rite for Children, Frisco, Texas
  - Texas Children's Hospital, Houston, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington
  - University of Washington, Seattle, Washington